CLINICAL TRIAL: NCT06559748
Title: A Multi-arm Randomized Controlled Trial of Transcranial Magnetic Theta-burst Stimulation in the Treatment of Functional Dyspepsia
Brief Title: A Trial of Transcranial Magnetic Stimulation in the Treatment of Functional Dyspepsia
Status: Temporarily not available | Type: Expanded Access
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0802
Record Dates: First submitted 2024-08-08; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-07

CONDITIONS: Functional Dysphonia
Keywords: Functional Dysphonia，Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: transcranial magnetic thetaburst stimulation （TBS） — TBS group: iTBS was administered to stimulate RMFC, 80-100% RMT, 10 times a course, twice a day, for a total of 5 days; Conventional drugs group: pantoprazole 40 mg orally once a day; itopride 50 mg orally three times a day; treatment for 4 weeks. （Standard medication regimen）
  Other Names: Conventional drugs

SUMMARY:
The goal of this clinical trial is to learn if theta burst stimulation (TBS), a form of Transcranial Magnetic Stimulation (TMS), can treat functional dyspepsia (FD) and compare its effectiveness against conventional drug treatments in patients diagnosed with FD. The main questions it aims to answer are:

Does TBS improve FD-related symptoms and associated mental health conditions such as anxiety and depression? How does the effectiveness of TBS compare to conventional drug treatments for FD?

Researchers will compare TBS treatment, sham TBS treatment, and conventional drug treatment to see if TBS is effective in treating FD. Participants will:

Undergo TBS or sham TBS treatment, or take conventional medications as prescribed.

Have their FD symptoms, anxiety, and depression levels assessed before and after the treatment.

Be evaluated at various intervals (Day 3, Month 1, Month 3, Month 6) for symptom improvement and side effects.

Participants are adults aged 18-70, diagnosed with FD, and willing to participate in this study. They will be randomly assigned to one of the three groups: TBS, sham TBS, or conventional drug treatment, with an equal number of participants in each group.

The study will be conducted over two years, from November 1, 2023, to October 31, 2025, at the Second Affiliated Hospital of Zhejiang University School of Medicine.

DETAILED DESCRIPTION:
Background:

Functional dyspepsia (FD) is a prevalent gastrointestinal disorder characterized by upper abdominal discomfort, including symptoms such as pain, bloating, early satiety, belching, and nausea. The etiology of FD is multifactorial, with psychosocial factors playing a significant role in its development. Recent advances in understanding the brain-gut axis have highlighted the potential of non-invasive neuromodulation techniques, such as Transcranial Magnetic Stimulation (TMS), to modulate brain activity and alleviate FD symptoms.

TMS, particularly theta burst stimulation (TBS), has shown promise in treating various neurological and psychiatric disorders. This study aims to explore the efficacy of TBS in improving both gastrointestinal symptoms and associated psychological symptoms in patients with FD, providing a novel therapeutic option for this challenging condition.

Objective:

The primary objective of this study is to compare the efficacy of TBS, sham TBS, and conventional pharmacological treatments in alleviating the symptoms of functional dyspepsia. The study seeks to determine whether TBS can offer superior symptom relief compared to standard treatment methods.

Study Design:

This is a single-center, randomized controlled clinical trial with 2 parallel arms: TBS treatment, and conventional drug therapy. Participants will be randomly assigned to one of the 2 groups in a 1:1 ratio. The study will be conducted over two years, from November 1, 2023, to October 31, 2025.

Intervention:

* TBS Group: Participants will receive iTBS stimulation of the right medial frontal cortex (RMFC) at 80-100% of their resting motor threshold (RMT), with 10 sessions per course, administered twice daily for five days.
* Conventional Drug Group:Participants will receive pantoprazole (40 mg orally once daily) and itopride (50 mg orally three times daily) for four weeks.

Participants:

The study will enroll 150 adult outpatients (aged 18-70 years) diagnosed with functional dyspepsia according to the Rome IV criteria. Participants will be screened based on specific inclusion and exclusion criteria and will provide informed consent before enrollment.

Data Management and Statistical Analysis:

All data will be collected and analyzed using SPSS 19.0 software. The analysis will include t-tests for normally distributed data and non-parametric tests for non-normally distributed data. The study will also employ multifactor ANOVA to assess the impact of various factors on treatment outcomes.

Ethical Considerations:

The study will be conducted in accordance with ethical standards, ensuring participant confidentiality and safety. Adverse events will be closely monitored and reported to relevant regulatory bodies.

This study aims to provide evidence for the clinical efficacy of TBS in treating FD, potentially offering a new therapeutic approach for managing brain-gut axis-related disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 years old, regardless of gender, outpatients.
2. Meets the Rome IV diagnostic criteria for functional dyspepsia in gastroenterology (2016 edition).
3. There are symptoms of postprandial fullness discomfort, early satiety discomfort, mid-upper abdominal pain, and mid-upper abdominal burning discomfort, with at least one score (degree + frequency) ≥ 4 points; the total score is ≥ 10 points. Note: See the case report form for the scoring table.
4. Agree to participate in this clinical trial and sign the informed consent form.

Exclusion Criteria:

1. Those who suffer from organic gastrointestinal diseases such as reflux esophagitis, peptic ulcer, gastrointestinal tumors, etc., or who are suspected of having intestinal obstruction.
2. Patients with intracranial hypertension, epilepsy, severe heart disease, other serious physical diseases or cognitive dysfunction; pregnant and lactating women.
3. ALT and AST are greater than 1.5 times the normal value, total bilirubin exceeds 1.5 times the upper limit of the normal value, and creatinine exceeds the upper limit of the normal value;
4. Suspected or confirmed history of drug or alcohol abuse;

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult